CLINICAL TRIAL: NCT06936722
Title: Comparison of McKenzie Protocol and ELDOA in Teachers With Non-Specific Neck Pain
Brief Title: McKenzie and ELDOA Comparison in Non-Specific Neck Pain Teachers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/ Umul Baneen 02003
Record Dates: First submitted 2025-04-14; First posted 2025-04-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Non Specific Neck Pain
Keywords: McKenzie Protocol for Neck Pain; ELDOA for Neck Pain; Pain; disability
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELDOA + Conventional PT (Experimental): ELDOA, the protocol consists of 4 positions. Each position is maintained for 1 min with constant correction of posture throughout with 2 to 4 min rest within each position. The Exercise was performed in 10 to 25 mins. 4 positions of ELDOA are Decoarctation of C0/C1/C2, Decoarctation of C4/C5, Decoarctation of C5/C6, Decoarctation of C6/C7. All positions are attained in lying.
  Hot pack 2. isometric strengthening exercises (Neck Flexion, Extension and Lateral Flexion) in 3x5 sets with 5 sec hold.
  Interventions: Other: ELDOA + Conventional PT
- McKenzie Protocol + Conventional PT (Active Comparator): Extension Dysfunction Retraction Retraction with patient overpressure Retraction with therapist overpressure Retraction with extension
  Lateral Flexion Dysfunction
  Lateral flexion:
  Lateral flexion with patient overpressure Lateral flexion therapist overpressure
  Rotation Dysfunction Rotation Rotation with patient overpressure
  Hot pack, isometric strengthening exercises (Neck Flexion, Extension and Lateral Flexion) in 3x5 sets with 5 sec hold Rotation with therapist overpressure
  Interventions: Other: McKenzie Protocol + Conventional PT

INTERVENTIONS:
Other: ELDOA + Conventional PT — ELDOA, the protocol consists of 4 positions. Each position is maintained for 1 min with constant correction of posture throughout with 2 to 4 min rest within each position. The Exercise was performed in 10 to 25 mins. 4 positions of ELDOA are Decoarctation of C0/C1/C2, Decoarctation of C4/C5, Decoarctation of C5/C6, Decoarctation of C6/C7. All positions are attained in lying.
  Hot pack 2. isometric strengthening exercises (Neck Flexion, Extension and Lateral Flexion) in 3x5 sets with 5 sec hold.
  Arms: ELDOA + Conventional PT
Other: McKenzie Protocol + Conventional PT — Extension Dysfunction Retraction Retraction with patient overpressure Retraction with therapist overpressure Retraction with extension Lateral Flexion Dysfunction Lateral flexion: Lateral flexion with patient overpressure Lateral flexion therapist overpressure Rotation Dysfunction Rotation Rotation with patient overpressure Hot pack, isometric strengthening exercises (Neck Flexion, Extension and Lateral Flexion) in 3x5 sets with 5 sec hold Rotation with therapist overpressure
  Arms: McKenzie Protocol + Conventional PT

SUMMARY:
The aim of this study is to compare the effectiveness of McKenzie Protocol and ELDOA on severity of pain, on the range of motion and disability level of teachers with Non-Specific neck pain.

DETAILED DESCRIPTION:
Neck pain, a common musculoskeletal condition and a common problem of the society, is "a pain originating from musculoskeletal tissue in the region from the Occiput to the First Thoracic Vertebrae". Approximately 2/3 of the population around Globe is affected by Neck Pain as it is the 4th leading cause of disability around the world. Several research has shown prevalence ranging between 14.2% to 71%, with increased frequency in females and middle-aged adults. Risk factors related to neck pain generally constitute trauma or sports related injuries, poor work environment and psychological issues. This common problem can further be categorized based on duration i.e. Acute (for less than 6 weeks), Sub Acute (for less than 3 months) and Chronic (For more than 3 months). Based on severity, it is further sub-divided into 3 categories (Mild, Moderate and Severe). Based on etiology it has 2 types, (Mechanical and Neuropathic) Non-Specific Neck pain (NNP), a broader term used, is a common appearance of Neck Pain elaborated as Pain without any defined cause. It can either be a Mechanical or a Postural complication. Non-Specific Neck pain can be diagnosed from the history of individual along with physical examination. Non-Specific Neck Pain responds to conservative management, but the recent Literature suggests that Exercise therapy is quite effective in treatment of Non-specific Neck Pain (NNP). Techniques include Exercise therapy, Manual therapy, Traction, Electrotherapeutic modalities, Stretching, Massage, Release Techniques (ARTs) which are effective not only for reducing Pain but also for improving Cervical Ranges and functional capacity of Individuals.

Teaching is considered among those Professions where Incidence of Neck pain is at its peak, a recent Literature suggest that Prevalence of Neck pain is 68.9% in teachers. Occupational Complications i.e. Long-standing hours, Faulty postures, Excessive use of electronic devices and Black boards are the major risk factors for teachers in developing Musculoskeletal Conditions, with an incidence of 40% to 95%.

McKenzie Protocol is an interventional approach used in the broader term of Exercise Therapy. A Literature published in International Journal of Physiotherapy and Research by researchers of Cairo University, Egypt showed that McKenzie Protocol is very effective for the treatment of Non-specific Spinal Pain. This technique encourages active patient involvement in decreasing pain which as a result increases the functional abilities of individuals. The Technique of Neck Retraction is very beneficial for increasing Cervical Ranges, improving Posture and relieving Neck pain. McKenzie Protocol is a very effective technique for preventing re-occurrence of Pain.

ELDOA an abbreviation used for a French acronym Elongation Longitudinaux avec Decoaption Osteo-Articulaire is a term described by Guy Voyer in 1979 as an active Traction technique used for stretching of Fascia and increasing Spacing of Spinal joints. Literature backs the claim that ELDOA is an effective technique used to decrease pain and increasing Muscle length. This technique release compression from the Facet joints which in return increase circulation and improves tone that helps in Pain reduction and Range improvement.

Neck Pain frequently affects teachers due to Occupational habits. According to the Global Burden of Disease (GBD) Study, neck pain is the second leading cause of years lived with disability (YLD) for adults, 50% - 75% of people do not recover from an acute episode and experience recurrent neck pain in the next 1 to 5 years. Approximately 68% of people develop persistent and chronic neck pain. A Meta-analysis focusing on the McKenzie Protocol indicated its efficacy in managing moderate to severe neck pain, relative to mild cases. Various studies have explored the individual effects of McKenzie and ELDOA techniques on Neck pain. However, no one has specifically investigated which protocol is more effective across different severity levels.

ELIGIBILITY:
Inclusion Criteria:

* Normal BMI
* Neck Pain on NPRS (Mild 1-3, Moderate 4-6, Severe 7-10)
* Working Hour: At least 30 hrs. per week.
* Teaching Experience: More than 12 months

Exclusion Criteria:

* No Neurological Condition (+ve Spurling Test, +ve Compression test, +ve Distraction Test)
* No Other Musculoskeletal Condition. (Osteoporosis, Arthritis, TrPs)
* No Spinal Deformity. (Scoliosis, Forward Head)
* No Surgery (Spinal Surgery, Fracture)
* No Cervical Tumor
* No complaints about Dizziness, Migraine, Cervicogenic headache (+ve Flexion Rotation test)

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Range of motion (Goniometer) | 3 weeks
  It is the most common instrument used to measure the range of motion of joints across the whole body. Normal ranges of cervical spine are Flexion approximately 80°, Extension 50°, Lateral bending 45° on either side and Rotation approximately 80°. Its Reliability (ICC = 0.82) and Validity (Correlations 0.97-0.98)
Numeric Pain Rating Scale NPRS | 3 weeks
  The NPRS is an eleven-point pain impression scale: the patient rates pain from 0 (no aggravation) to 10 (most exceedingly terrible possible pain). Mild 1-3, Moderate 4-6, Severe 7-10. Numeric Pain Rating Scale (NPRS), which was used to survey respondents' impression of the degree of pain that they felt. It is an outcome measure that is a unidimensional measure of pain intensity in adults. It is considered a more objective and Numeric version of Visual Analogue Scale.
Neck Disability Index or NDI | 3 weeks
  It has sufficient support and usefulness to retain its status as the most used self-report disability measure for neck pain. 0 to 4 = no disability, 5 to 14 = mild, 15 to 24 = moderate, 25 to 34 = severe, above 34 = complete. It has ten sections with each section carrying 5 marks.

CONTACTS AND LOCATIONS:
Overall Officials: Maria khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Yusra Medical and Dental College, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No